CLINICAL TRIAL: NCT00450944
Title: A Phase I Study of Combination Therapy With Anti-CD19 and Anti-CD22 Immunotoxins (Combotox) in Adults With Refractory/Relapse Acute Lymphoblastic Leukemia
Brief Title: Anti-CD19 and Anti-CD22 Immunotoxins in Treating Patients With Refractory or Relapsed B-Cell Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-536; P30CA013330 (NIH); AECM-CCI-2005-536; AECM-CCI-05-428; AECM-MMC-05-10-265C; NCT00272298 (obsolete NCT alias)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Leukemia
Keywords: B-cell adult acute lymphoblastic leukemia; recurrent adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — combotox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: Yes

ARMS (1):
- Combination Therapy with Immunotoxins Imtox 19 Plus Imtox 22 (Experimental)
  Interventions: Biological: deglycosylated ricin A chain-conjugated anti-CD19/anti-CD22 immunotoxins

INTERVENTIONS:
Biological: deglycosylated ricin A chain-conjugated anti-CD19/anti-CD22 immunotoxins

SUMMARY:
RATIONALE: Immunotoxins, such as anti-CD19 and anti-CD22, can find cancer cells that express CD19 and CD22 and kill them without harming normal cells. This may be an effective treatment for B-cell acute lymphoblastic leukemia.

PURPOSE: This phase I trial is studying the side effects and best dose of anti-CD19 and anti-CD22 immunotoxins in treating patients with refractory or relapsed B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of deglycosylated ricin A chain-conjugated anti-CD19 and anti-CD22 immunotoxins (Combotox) in patients with refractory or relapsed B-cell acute lymphoblastic leukemia.
* Determine the toxicity of Combotox in these patients.
* Determine the pharmacokinetic (PK) profile of Combotox in these patients.
* Determine any antitumor activity of Combotox, in terms of the percentage of blasts in bone marrow and peripheral blood.
* Determine the levels of human antimouse and human anti-dgA antibodies in patients treated with Combotox.
* Determine if there is a correlation between PK parameters and toxicity of Combotox in these patients.
* Determine if the expression of the CD19 and CD22 cell surface antigens is affected by Combotox.

OUTLINE: This is a dose-escalation study.

Patients receive deglycosylated ricin A chain-conjugated anti-CD19 and anti-CD22 immunotoxins (Combotox) IV over 4 hours on days 1, 3, and 5 in the absence of disease progression or unacceptable toxicity.

Cohorts of patients receive escalating doses of Combotox until the maximum tolerated dose is determined.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adult acute lymphoblastic leukemia

  * B-cell lineage
* Refractory or relapsed disease based on a bone marrow/peripheral blood examination, cytogenetic studies, or polymerase chain reaction amplification

  * Disease refractory to conventional therapy and other therapies of higher priority
* At least 50% of the blasts (in bone marrow or peripheral blood) expressing CD19 and/or CD22 by flow cytometry

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 2 months
* Creatinine < 1.5 times normal
* Bilirubin < 1.5 times normal
* ALT or AST < 2.5 times normal

PRIOR CONCURRENT THERAPY:

* Prior chemotherapy, biologic therapy, and/or radiotherapy allowed

Ages: 17 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-02-22 (Actual); Primary Completion 2008-10-27 (Actual); Study Completion 2010-04-01 (Actual)

PRIMARY OUTCOMES:
Optimum dose of deglycosylated ricin A chain-conjugated anti-CD19 and anti-CD22 immunotoxins (Combotox)
Efficacy of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amit Verma, MD, Study Chair — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York, United States